CLINICAL TRIAL: NCT04006860
Title: A Single-center, Open-label, Randomized, Two-period Crossover Food-effect Study of SHC014748M in Healthy Subjects
Brief Title: A Food-Effect Study of SHC014748M in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHC014-I-02
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHC014748M: Fast + Fed (Experimental): Participants will receive a single oral dose of SHC014748M capsules in fasted condition on Day 1 of treatment period 1 followed by a single oral dose of SHC014748M capsules in fed condition on Day 8 of treatment period 2.
  Interventions: Drug: SHC014748M Capsules
- SHC014748M: Fed + Fast (Experimental): Participants will receive a single oral dose of SHC014748M capsules in fed condition on Day 1 of treatment period 1 followed by a single oral dose of SHC014748M capsules in fasted condition on Day 8 of treatment period 2.
  Interventions: Drug: SHC014748M Capsules

INTERVENTIONS:
Drug: SHC014748M Capsules — SHC014748M Capsules: 200mg

SUMMARY:
The primary objective of this study is to determine the effect of food in healthy participants on the bioavailability of SHC014748M Capsules following single dose administration with and without a meal.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, two-period, crossover PK food effect study of SHC014748M Capsules administered orally at 200 mg.

For each of 2 study periods, subjects will be admitted to the clinical research unit on the day before dosing and fast overnight (approximately 10 hours). On the morning of dosing for each of the 2 study periods, subjects will receive a single oral dose of 200 mg SHC014748M Capsules in either the fasted or fed state. Subjects will remain at the clinical research unit for at least 72 hours after administration of study drug for collection of serial blood samples for pharmacokinetic (PK) analysis and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male subject,18-45 years of age.

  2. BMI between 19 and 26; Weight between 50 and 80 kg.

  3. Healthy medical examination ,various laboratory inspection indicators normal, or the abnormal signs have no clinical significance.

  4. Subjects (including their partners) who are willing to voluntarily take effective contraceptive measures from screening to 6 months after the last dose.

  5. Sign the informed consent form before the study and fully understand the study content, process and possible adverse reactions.

Exclusion Criteria:

* 1. Nervous system, respiratory system, cardiovascular system, digestive system, blood and lymphatic system, endocrine system, musculoskeletal system, etc. are abnormal and have clinical significance as determined by investigator.

  2. History of severe allergy/hypersensitivity or or ongoing allergy/hypersensitivity.

  3. Addicted to smoking and drinking in 3 months before the trial.

  4. Hemorrhage over 200mL , receive blood transfusions or use blood products in 3 months before the trial.

  5. Other conditions not suitable for trial, by judgement of investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
AUC(0-t) | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of the area under the plasma concentration-time curve from zero to last measurable concentration.
AUC(0-∞) | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of the area under the plasma concentration-time curve from zero to infinity
Cmax | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of maximum plasma concentration

SECONDARY OUTCOMES:
tmax | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of time to Cmax
AUC[%Extrap obs] | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of AUC[%Extrap obs],the rate of AUC(t-∞) to AUC
t l/2 | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of Terminal half life
λz | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of terminal rate constant
CL/F | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of apparent plasma clearance
Vz/F | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of apparent volume of distribution
MRT | 72 hours
  Pharmacokinetic of SHC014748M Capsules by assessment of Mean Residence Time

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No